CLINICAL TRIAL: NCT04731870
Title: Exploring Vaccine Confidence and Uptake of Potential COVID-19 Vaccines Among a Cross-section of US Healthcare Providers and Key At-risk Subgroups in the Rural South
Brief Title: Exploring Vaccine Confidence and Uptake of Potential COVID-19 Vaccines
Status: Completed | Type: Observational
Sponsor: East Carolina University (Other)
Responsible Party: Sponsor
Other Study IDs: 60622
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-03

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nurses/Doctors: Covid-19 vaccine confidence and recommendation practices of nurses/doctors
  Interventions: Other: Survey research
- Minority populations living in rural south: Covid-19 vaccine confidence and uptake of key at-risk subgroups and tailored Covid-10 vaccine messaging for at-risk subgroups.
  Interventions: Other: Survey research

INTERVENTIONS:
Other: Survey research — This is not an intervention study. It involves social science research of surveys and focus groups.

SUMMARY:
The COVID-19 pandemic has highlighted deleterious US health inequities. Specifically, African Americans, Latinos, and Native Americans have and continue to shoulder a greater burden of COVID-19 infections and deaths in the US. In addition to existing racial and ethnic disparities are rural health and regional disparities. Given the disproportionate impact of disease in US communities of color and also in rural and southern regions of the US, there is no doubt that these at-risk subgroups will continue to experience higher rates of coronavirus-related mortality as well as other long-term health outcomes as compared to other US populations.

It is unknown how healthcare providers and other key at-risk subgroups within the US will receive COVID-19 vaccines. For success in immunizations, the US will need to reach their most at-risk and vulnerable populations. In addition to at-risk populations, a successful immunization strategy will involve engaging providers to support clear, consistent, and strong vaccine recommendation. It is critical to build vaccine trust, confidence, and overall acceptance of COVID-19 vaccines among healthcare providers and key at-risk subgroups, especially given the accelerated production timeline of these vaccines. Likewise, tailored vaccine messaging for key subgroups is vital in achieving vaccine confidence and trust.

The proposed study will explore perceptions, confidence, trust, and uptake of potential COVID-19 vaccines among healthcare providers (nurses and doctors) and key at-risk population subgroups (minority populations living in the rural south) and will develop and test vaccine messaging that boosts vaccine confidence and trust among these key at-risk subgroups.

DETAILED DESCRIPTION:
Study objectives are as follows: Objective 1: To assess COVID-19 perceptions, COVID-19 vaccine confidence, projected vaccine recommendation practices, and trust in the health system and public health authorities among a cross-section of healthcare providers in the US (nurses and physicians); Objective 2: To assess COVID-19 perceptions, COVID-19 vaccine confidence, projected vaccine uptake, and trust in the health system, in healthcare providers, and in public health authorities among key at-risk subgroups in the US (minority populations living in the rural south); and Objective 3: To develop, tailor, and test COVID-19 vaccine messaging to boost vaccine confidence and trust, and COVID-19 preventive behavior, among at-risk subgroups in the US (minority populations living in the rural south). Perceptions, confidence, uptake, and trust in potential COVID-19 vaccines will be assessed among four identified and distinct groups via a quantitative and electronic survey and qualitative focus groups with key at-risk subgroups will be utilized to develop, tailor, and test COVID-19 vaccine messaging for at-risk subgroups.

This study will: 1) provide important national-level data regarding healthcare provider vaccine perceptions, confidence, trust, and projected vaccine recommendation practices for COVID-19, 2) ascertain vaccine perceptions, confidence, trust, and projected uptake of potential COVID-19 vaccines among at-risk populations in the US, and 3) develop tailored messaging for at-risk populations that can be used to boost vaccine confidence and trust, and preventive behaviors, among these high-risk groups in the coming years. This study will help to inform a larger coordinated national promotion strategy and campaign that can work to effectively communicate with the public about potential COVID-19 vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Nurses (at least 50% from the south),
2. Primary Care/Family Physicians (at least 50% from the south),
3. Rural, low-income, minority men and women living in the south (income of $25K per year or less and 70% of respondents will be Black, Latina, or Native American) and
4. Urban, low-income minority men and women living in the south (income of $25K per year or less and 70% of respondents will be Black, Latina, or Native American).

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Objectives 1 and 2 will be met by administering an electronic quantitative survey among the following four distinct groups: 1) Nurses (at least 50% from the south), 2) Primary Care/Family Physicians (at least 50% from the south), 3) Rural, low-income, minority men and women living in the south (income of $25K per year or less and 70% of respondents will be Black, Latina, or Native American) and 4) Urban, low-income minority men and women living in the south (income of $25K per year or less and 70% of respondents will be Black, Latina, or Native American). Each group will contain at least 150 subjects for a total of 600 participants.
Sampling Method: Non-Probability Sample
Enrollment: 632 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Covid-19 vaccine confidence (survey to be developed by study team) | year 1
  Confidence in the Covid-19 vaccine efficacy and safety among a cross-section of healthcare providers and key at-risk subgroups in the US
Covid-19 vaccine messaging (messages to be developed by study team & focus group participants) | year 2
  COVID-19 vaccine messaging (e.g. one or two sentences of culturally appropriate messages) that can be used to boost vaccine confidence and trust, and COVID-19 preventive behavior, among at-risk subgroups in the US (minority populations living in the rural south).
Covid-19 vaccine uptake (survey to be developed by study team) | year 1
  COVID-19 vaccine uptake or projected uptake among a cross-section of healthcare providers and key at-risk subgroups in the US
Covid-19 vaccine trust (survey to be developed by study team) | year 1
  COVID-19 vaccine trust in the health system and public health authorities a cross-section of healthcare providers and key at-risk subgroups in the US
Covid-19 vaccine recommendation practices (survey to be developed by study team) | year 1
  COVID-19 vaccine recommendation practices among a cross-section of healthcare providers in the US

CONTACTS AND LOCATIONS:
Overall Officials: Becky Welch, CPA, Study Chair — Assistant Vice Chancellor for Research Administration & Finance
Locations (1):
- Carol Belk Building, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No